CLINICAL TRIAL: NCT06149806
Title: National Registry of Adult Heart Failure Patients With Complex Congenital Heart Disease: Systemic Right Ventricle and Single Ventricle Treated With Sacubitril/Valsartan
Acronym: ISACC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.003
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Complex Congenital Heart Disease
MeSH Terms: interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- efficacy and tolerability of Sacubitril/Valsartan: efficacy and tolerability of Sacubitril/Valsartan in the treatment of chronic heart failure on complex congenital cardiopathy
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet [Entresto]

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet [Entresto] — efficacy and tolerability of Sacubitril/Valsartan in the treatment of chronic heart failure on complex congenital cardiopathy

SUMMARY:
Heart failure in adults with congenital heart disease is a major cause of morbidity and mortality. Patients with systemic right ventricle (SRV) and single ventricle (SV) are particularly at risk1, 2, 3.

There are no specific recommendations for the management of heart failure in adults with congenital heart disease, whose management is based on "general cardiology" recommendations4,5.

Sacubitril/Valsartan is validated as a treatment for heart failure in adults with acquired pathological left ventricular dysfunction (left ventricular ejection fraction (LVEF) < 40%, New York Heart Association (NYHA) functional class II and III despite optimal heart failure therapy)7. Although this molecule is used in current practice in patients with congenital heart disease, published data are limited 6-10.

The aim of our work is to describe the efficacy and tolerability of Sacubitril/Valsartan in the treatment of chronic heart failure on VDS and VU through an observational, prospective, multicenter registry.

The latest heart failure treatment guidelines, updated in 202111, recommend the addition of type 2 sodium-glucose co-transport inhibitors in heart failure patients with impaired ejection fraction (class IA recommendation). Two molecules are used in current practice: dapagliflozin and empagliflozin, at a single dosage of 10 mg/day.

We will also be collecting data on the efficacy and safety of iSGLT2. It should be noted that, for practical reasons, there may be a delay between the end of the 1st study period (ISACC1) of one year and the start of the 2nd study period (ISACC2).

Follow-up examinations carried out during the study period will not differ from those currently recommended in current practice5.

ELIGIBILITY:
Inclusion Criteria:

* - Patients ≥ 18 years of age
* Congenital heart disease with systemic right ventricle (D-TGV after atrial switch (Mustard or Senning surgery) or double mismatch), single ventricle of right or left morphology
* Systemic ventricular ejection fraction ≤ 40% (on cardiac magnetic resonance imaging (MRI) less than 12 months old).

In case of contraindication to MRI, LVEF ≤ 40% if systemic left ventricle or surface shortening fraction ≤ 35% if VDS12 (examination less than 12 months old).

* NYHA II or III
* On optimal heart failure therapy: ACE inhibitor or ARB2 for ≥ 4 weeks, at maximum tolerated dose. Whether or not combined with beta-blockers and maximum-tolerated-dose mineralocorticoid receptor antagonists.
* Cardiopulmonary exercise test (CPET) within the last 12 months

Exclusion Criteria:

* - Other congenital heart disease
* Inability to perform CPETH
* Immuno-allergic reaction, history of angioedema on ACE inhibitors or ARB2 inhibitors
* Symptomatic arterial hypotension or BPs < 100 mHg
* Renal insufficiency (GFR <30 mL/min/m²), hyperkalemia > 5.4 mmol/l, severe hepatic insufficiency (Child-Pugh Class C)
* Pregnancy or breast-feeding
* Opposition to use of patient data
* Type 1 diabetes if on iSGLT2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Congenital heart disease with systemic right ventricle or unique ventricle.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To describe the 12-month (± 2 months) evolution of functional capacity during CPETH in adult heart failure patients with dysfunctional VDS or VU treated with Sacubitril/Valsartan. | 12 months
  Comparison of peak VO2 during CPETH before introduction of Sacubitril/Valsartan and at 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided